CLINICAL TRIAL: NCT05448911
Title: The Role of Intraoperative Navigation-assisted Channel Screw Technique in the Treatment of Pelvic Fractures: A Multicenter, Prospective, Randomized, Controlled Study
Brief Title: The Role of Intraoperative Navigation-assisted Channel Screw Technique in the Treatment of Pelvic Fractures
Acronym: INCST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2020-011
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-06

CONDITIONS: Pelvic Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): It uses minimally invasive small incisions, physiological access to the pelvis, and hollow screws for Pelvic and Acetabular fractures
  Interventions: Procedure: Intraoperative navigation combined with Catheter screw technique
- Control Group (Other): This approach typically requires extensive surgical exposure and large-scale soft-tissue dissection, which quickly leads to some serious complications, including increased rates of infection, poor wound healing, increased damage to large vessels or nerves, and heterotopic ossification
  Interventions: Procedure: Open reduction and internal fixation with steel plate

INTERVENTIONS:
Procedure: Intraoperative navigation combined with Catheter screw technique — It uses minimally invasive small incisions, physiological access to the pelvis, and hollow screws for Pelvic and Acetabular fractures
  Arms: Experimental group
Procedure: Open reduction and internal fixation with steel plate — Open reduction and plate internal fixation is the most commonly used method to treat pelvic fracture, which can achieve anatomical reduction and rigid fixation. However, this method requires extensive dissection of the surrounding soft-tissue fracture and is invasive
  Arms: Control Group

SUMMARY:
This was a multicenter, prospective, randomized, controlled study. Patients with pelvic fractures (Tile B and c) were recruited from the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an Red Society Hospital and Xi'an 521 hospital, the patients were randomly divided into two groups according to the Order of admission: Experimental Group (intraoperative navigation combined with channel screw technique) and Control Group (open reduction and plate internal fixation) , the difference of operative effect between the two groups was compared by fracture reduction, channel screw position, operative time, fluoroscopy frequency, hospitalization time, hospitalization cost, recovery time and Mayo Score. Use Access 2003 to build a database and store data; use SPSS 21.0. 0 Software for statistical analysis. The entire process required the development of a standardized staff manual, and all were subject to rigorous training and examination in order to participate in the pilot, and the investigation process was supervised by the project leader.

DETAILED DESCRIPTION:
With the rapid development of the transportation industry and construction industry, pelvic fractures caused by high-energy injuries are increasing year by year, accounting for about 3% -5% of total body fractures. This disease seriously endangers the lives of patients. Once it occurs, the mortality and disability rate are high. Finding the appropriate treatment has been the direction explored by orthopedic surgeons . Undisplaced pelvic fractures can usually be treated conservatively, which has the advantages of low cost and minor trauma, but heavily displaced fractures often require surgery due to the destruction of pelvic stability structures. Conservative treatment cannot achieve functional reduction or even anatomical reduction (Fig. Traditional open reduction and internal fixation with steel plate is the mainstream treatment at present. Still, this method usually requires extensive surgical exposure and massive dissection of soft tissue, which quickly causes some severe complications, including increased infection rate, poor wound healing, increased macrovascular or nerve injury, and heterotopic ossification . At the same time, with the arrival of an aging society, there are more and more pelvic fractures in the elderly in clinical practice, and the treatment faces many challenges. First, the elderly have a poor physical conditions, are primarily associated with medical diseases of varying severity, and have poor tolerance to surgery. Second, with different degrees of decreased bone conditions, some patients with severe osteoporosis have fractures that are difficult to reduce and effectively fix. Their treatment far exceeds the choice between conservative treatment and surgical treatment, requiring multidisciplinary teamwork, including orthopedics, geriatrics, endocrinology, pain, and rehabilitation physiotherapy. The principle of treatment for elderly patients with a pelvic fracture is as follows: while the fixation is as strong as possible, minimally invasive fixation should be adopted as far as possible to reduce the surgical blow and related complications. Therefore, the minimally invasive channel screw technique has become a hot spot in the treatment of pelvic fractures.

In recent years, the minimally invasive channel screw technique has been gradually paid attention to by clinicians. It mainly uses a minimally invasive small incision, uses the physiological channel of the pelvis, and uses cannulated screws to fix pelvic and acetabular fractures. This technique provides a reliable and stable fixation of the pelvic acetabulum, which is equivalent to or superior to other existing internal fixation techniques such as plates from a biomechanical point of view, can achieve the effect of open reduction and internal fixation and can avoid complications such as more bleeding and extensive soft tissue dissection caused by open surgery, which will become the most popular method for the treatment of pelvic acetabular fractures.

The project group previously tried the channel screw technique for the treatment of pelvic fractures and found that although this method has the advantages of minimally invasive and rapid recovery, it still has the following problems: due to the small incision, it cannot fully expose the visual field and is easy to damage the peripheral blood vessels and nerves. Continuous fluoroscopy under the C-arm is required, and the radiation dose received by patients and physicians is large; for the technical and empirical requirements of physicians, the learning curve of young physicians is high. General anesthesia is used during the operation, which increases the risk of removal of the endotracheal tube if the operation time is high. The development and popularization of intraoperative navigation technology provide the possibility to solve the above problems.

Navigation technology is widely used in many fields such as transportation, exploration, military, and exploration. With the continuous development of computer technology, especially the rapid progress of computer graphics technology, a new field of computer-assisted surgery (CAS) has emerged, and computer-assisted navigation system (CANS) is an important part of it. The computer-assisted surgical navigation system is a combination of spatial three-dimensional stereotactic technology, modern imaging diagnostic technology, computer image processing technology, three-dimensional visualization technology, and minimally invasive surgical techniques. It uses signal transmission, transmission, and reception transmitters to calculate the data of each position point through a computer to obtain the required various curves and angles so that the various parameters of the intangible and virtual human body are converted into direct animated images while the position of surgical instruments is displayed in real-time on the surgical images, and the doctor can understand the relationship between the position of instruments and anatomical structures at any time so that the surgical operation becomes safer, more accurate and less invasive.

The current application of navigation technology in orthopedics is mainly focused on spinal surgery, which is less used in the field of trauma. Due to the special anatomy of the spine and spinal cord, the high accuracy and safety of surgery are the first considerations. In 1995, Nolte implemented the world's first lumbar pedicle screw internal fixation surgery using a computer-assisted minimally invasive navigation surgical system, which began the use of navigation technology in spinal surgery, and Nolte et al. found that the accuracy of the photoelectric spinal navigation system could reach 1-1.7 mm, and image-guided technology allowed surgeons to clearly understand the spinal anatomy and the pedicle screw needle insertion point and needle insertion direction, and fixed pedicle screws in the correct position of the vertebral body by real-time tracking to improve the surgical accuracy. Channel screw therapy for pelvic fractures is a difficult surgery in the field of trauma. Navigation is used during screw placement. The specific position of the guide needle can be determined according to the real-time three-dimensional picture displayed by the system. The direction of the real guide needle can be corrected by adjusting the direction of the virtual guide needle in time during surgery, providing a safety guarantee for screw placement .

In this study, the patients with pelvic fractures (Tile B and C) admitted to the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an Red Cross Hospital, and Xi'an 521 Hospital were used as the cohort study basis, intraoperative navigation combined with channel screw technique was used as the experimental group, and open reduction and internal fixation with steel plate were used as the control group. Through intraoperative evaluation and postoperative follow-up, the surgical effects were compared between the two groups. To explore the significance of intraoperative navigation assisted channel screw technology in the treatment of pelvic fracture, expect that this treatment can reduce the number of fluoroscopies, shorten the operation time, improve postoperative satisfaction of patients, reduce the length of hospital stay and reduce medical costs, and finally this treatment method can be popularized and applied.

ELIGIBILITY:
Inclusion criteria

1. inpatients diagnosed with unstable pelvic acetabular fractures (tile B, C);
2. sacroiliac joint dislocations and longitudinal sacral fractures that do not require sacral nerve or sacral canal decompression;
3. closed reduction to functional reduction criteria before posterior pelvic ring. Exclusion Criteria

1)stable posterior pelvic ring injury (Tile A type); 2)preoperative closed reduction to achieve functional reduction; 3)patients with severe osteoporosis; 4)heart, liver, kidney, and other essential organ lesions cannot tolerate surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic change | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 month
  fracture displacement < 4 mm was excellent, 4-10 mm was good, 10-20 mm was fair, and > 20 mm was poor.

SECONDARY OUTCOMES:
screw position | follow-up of 3 months, 6 months and 12 months
  Class I, safe implantation, the screw was completely in the cancellous bone; Class II, safe implantation, the screw contacted the cortical structure ; Class III, wrong implantation, the screw penetrated the cortical bone.
pubic ramus screws | follow-up of 3 months, 6 months and 12 months
  grade 0, no penetration of the bone cortex; grade 1, penetration of the bone cortex screw length < 2 mm; grade 2, penetration of the bone cortex screw length 2-4 mm; grade 3, penetration of the bone cortex screw length > 4 mm.
VAS scores VAS scores | follow-up of 3 months, 6 months and 12 months
  Evaluation of postoperative pain
The length of hospital stay | follow-up of 3 months, 6 months and 12 months
  The total length of stay of the patient in the hospital
Total cost of hospitalization | follow-up of 3 months, 6 months and 12 months
  Overall cost of hospitalization
Pelvic X-ray was taken to record the fracture healing, hip joint function | follow-up of 3 months, 6 months and 12 months
  X-ray evaluation of fracture healing